CLINICAL TRIAL: NCT03579134
Title: Evaluation of Patient Satisfaction and Adaptation After Elevation of Vertical Dimension of Occlusion in Patients With Compensated Tooth Surface Loss Using Partial Overlay Denture or Fixed Temporary Crowns
Brief Title: Satisfaction and Adaptation After Elevation of Vertical Dimension of Occlusion Using Overlay Denture or Fixed Crowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Elkammah, Principal inverstigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: amrelkammah
Record Dates: First submitted 2018-06-08; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- partial overlay denture (Experimental): removable partial denture with a metal extension over the remaining posterior teeth raising their height to the newly proposed vertical dimension and occlusal plane
  Interventions: Device: partial overlay denture
- fixed temporary crowns (Active Comparator): fixed crowns made from temporary material placed on the prepared posterior teeth to the new occlusal plane level elevating the vertical dimension to the newly proposed level
  Interventions: Other: fixed temporary crowns

INTERVENTIONS:
Device: partial overlay denture — removable appliance similar to a removable partial denture but with overlay occluslal rests covering the full occlusal surface of the remaining posterior teeth
  Arms: partial overlay denture
Other: fixed temporary crowns — fixed crowns made from temporary material placed to the newly altered vertical dimension
  Arms: fixed temporary crowns

SUMMARY:
Elevation of the vertical dimension of occlusion has always been a debatable issue specially using removable prosthesis. Fixed restorations have been a more predictable treatment modality in treating patients with tooth surface loss. A more conservative restoration, more retrievable, and cost effective option is proposed. Partial overlay dentures could provide a reversible and more conservative solution either by being used as a final restoration or teeth are provided with ceramic onlays instead of crowns.

DETAILED DESCRIPTION:
Tooth surface loss and its prevalence:

Tooth surface loss is a process that describes loss of hard tooth structure due to reasons other than caries, trauma, or developmental disorders. Lambrechts et al. in 1989 estimated that the physiological tooth surface loss per annum to be approximately between 20-38 micrometers.

More than the average amount of TSL could be described as pathological tooth surface loss. A systematic review of 186 prevalence studies reported an increase of tooth surface loss from 3% at the age of 20 to 17% at the age of 70. Another German study reported similar results.

Pathologic tooth surface loss:

Pathologic tooth surface loss can be classified into attrition, abrasion, erosion, and abfraction.

These factors in addition to overloaded teeth due to partial edentulism can cause loss in the vertical dimension of occlusion (non-compensated by alveolar bone) or loss of tooth substance with dento-alveolar growth preserving the vertical dimension but with unsatisfactory esthetics and sometimes dentine exposure and sensitivity. Vertical dimension of occlusion according to the glossary of prosthodontics is defined as the distance measured between two points when the occluding members are in contact.

Loss of vertical dimension:

Elevation of vertical dimension of occlusion has different modalities. The choice between the treatment options depends mainly on the extent of tooth surface loss (which can be quantified by different classification indices as the popular Smith and Knight classification and the more recent BEWE classification described by Bartlett at 2010), and the aesthetic needs of different patients.

Deciding to go for a restorative treatment can be subdivided into one of three lines which are:

* Altering position of the mandibular closure while maintaining the existing vertical dimension which can only be accomplished in teeth when no need to restore anterior teeth and the rest of the posterior teeth are sound. This concept is based on the different in position between the vertical dimension of occlusion and the centric relation.
* Increasing the vertical dimension of occlusion.
* axial tooth movement through orthodontic treatment of prosthodontic appliances inducing orthodontic forces.

Compensated and non-compensated tooth surface loss:

Tooth surface loss can be either compensated where the freeway space remains within the normal range due to overgrowth of the teeth with the alveolar bone into axial direction, and non-compensated tooth surface loss leading to loss of occlusal vertical dimension and increase in the average freeway space (2-3mm).

Need for esthetic and functional rehabilitation in addition to covering sensitive exposed dentine in both cases urges treatment.

While non-compensated tooth surface loss presents a more predictable and easier modalities of treatment where the freeway space exceeds the average of 2mm, so it is easy to quantify the amount needed to be raised; compensated tooth surface loss based on available studies reported establishment of a new postural position of the mandible and new interocclusal distance obtained even when violating the freeway space.

Based on the previous findings we decided to study alteration of the vertical dimension of occlusion in patients with compensated tooth surface loss.

One group temporized during adaptation period with partial overlay denture and the other using fixed temporary crowns on the new vertical dimension of occlusion. This new vertical dimension is determined according to a wax up where patients included require esthetic alteration between 2-5mm.

Different techniques of alteration of the vertical dimension of occlusion differed between fixed and removable prosthesis through temporization (adaptation period).

Removable prosthesis had the advantage of retrievability, while the fixed ones had the advantage of ensuring patient adherence while symptoms persist.

The investigator's subject groups are fully dentate or partially edentulous patients (free end or long bounded posterior) with at least a pair of occluding posterior teeth on each side. Subjects have moderate to severe tooth surface loss requiring elevation of vertical dimension of occlusion from 2-5mm.

Subjects will be restored using patial overlay denture or fixed temporary crowns.

Partial overlay denture is similar to temporary partial dentures with occlusal extension of teeth where the existing posterior teeth can reach the newly reorganized occlusal plane.

A systematic review conducted in Germany reported symptoms collected from different articles associated with elevation of the vertical dimension of occlusion. These symptoms included headache, tenderness in the masseter and temporalis muscle area upon palpation, clenching, grinding muscle and joint fatigue, soreness of teeth, cheek biting and difficulty in chewing and swallowing.

Studying the two different groups is intended to monitor whether or not these symptoms appear, severity of these symptoms, time taken for alleviation of these symptoms if it does and overall patient satisfaction. Adaptation period will be up to 3 month through which a weekly recall will be done to evaluate adaptation. Patients satisfaction is reported weekly until adaptation occurs or at the end of the time limit using OHIP questionnaire.

Fixed restorations has the benefit of comfort and adherence of the patient over removable options while it might need full crowning with less conservatism and more cost. The partial overlay denture as a removable prosthesis is also less comfortable for the patient but could be proposed as a retrievable, more conservative and a cheaper option.

ELIGIBILITY:
Inclusion Criteria:

* Patients fully dentate or partially edentulous with medium to severe tooth surface loss
* Minimum of one existing occluding pair of posterior teeth on each side (right and left).
* Patients were class 1 skeletal relation Patients requiring elevation 2-5mm.
* Patients having compensated tooth surface loss

Exclusion Criteria:

* Patients not having atleast 2 occluding pairs of posterior teeth.
* Skeletal class 2 and 3.
* Edentulous patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Assesment of patient satisfaction using OHIP-14 questionnaire | 3 months
  comfort of the patient and satisfaction regarding function, speech, esthetics are assesed using OHIP-14 questionnaire, and assesment will be using a Likert scale. The Likert Scale is a 5 or 7 point scale that offers a range of answer options - from one extreme attitude to another, like "extremely likely" to "not at all likely." Typically, they include a moderate or neutral midpoint.

SECONDARY OUTCOMES:
adaptation | 3 months
  absence of any appearing symptoms associated with elevating the vertical dimension of occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Amr H Elkammah, B.D.S, Principal Investigator — Cairo University; Ahmed E Fayyad, P.H.D, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: the use of a controlled access approach, using a transparent and robust system to review requests and provide secure data access, seeking consent for sharing IPD from participants with adequate assurance that patient privacy and confidentiality can be maintained; and establishing an approach to resource the sharing of IPD

REFERENCES:
- [Background] Abduo J. Safety of increasing vertical dimension of occlusion: a systematic review. Quintessence Int. 2012 May;43(5):369-80. PMID 22536588
- [Background] Beddis HP, Durey K, Alhilou A, Chan MF. The restorative management of the deep overbite. Br Dent J. 2014 Nov;217(9):509-15. doi: 10.1038/sj.bdj.2014.953. PMID 25377818
- [Background] Davies SJ, Gray RJ, Qualtrough AJ. Management of tooth surface loss. Br Dent J. 2002 Jan 12;192(1):11-6, 19-23. doi: 10.1038/sj.bdj.4801278. PMID 11852896
- [Background] Faigenblum M. Removable prostheses. Br Dent J. 1999 Mar 27;186(6):273-6. doi: 10.1038/sj.bdj.4800086. PMID 10230101
- [Background] Ibbetson R. Tooth surface loss. 9. Treatment planning. Br Dent J. 1999 Jun 12;186(11):552-8. doi: 10.1038/sj.bdj.4800167. No abstract available. PMID 10405470
- [Background] Lambrechts P, Braem M, Vuylsteke-Wauters M, Vanherle G. Quantitative in vivo wear of human enamel. J Dent Res. 1989 Dec;68(12):1752-4. doi: 10.1177/00220345890680120601. PMID 2600255
- [Background] Mehta SB, Banerji S, Millar BJ, Suarez-Feito JM. Current concepts on the management of tooth wear: part 2. Active restorative care 1: the management of localised tooth wear. Br Dent J. 2012 Jan 27;212(2):73-82. doi: 10.1038/sj.bdj.2012.48. PMID 22281629
- [Background] Carlsson GE, Ingervall B, Kocak G. Effect of increasing vertical dimension on the masticatory system in subjects with natural teeth. J Prosthet Dent. 1979 Mar;41(3):284-9. doi: 10.1016/0022-3913(79)90008-8. No abstract available. PMID 283228
- [Background] Gopi Chander N, Venkat R. An appraisal on increasing the occlusal vertical dimension in full occlusal rehabilitation and its outcome. J Indian Prosthodont Soc. 2011 Jun;11(2):77-81. doi: 10.1007/s13191-011-0066-9. Epub 2011 May 27. PMID 22654346